CLINICAL TRIAL: NCT04901364
Title: Sensitivity and Specificity Study of Risk Factors for Intraductal Papillary Mucinous Neoplasms Degeneration at the Nancy CHRU (IPMN)
Brief Title: Study of Risk Factors for Intraductal Papillary Mucinous Neoplasms Degeneration at the Nancy CHRU (IPMN)
Acronym: IPMN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Jean-Baptiste CHEVAUX, PH, Central Hospital, Nancy, France
Other Study IDs: 2021PI064
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Study of Risk Factors for IPMNs Degeneration at the Nancy CHRU
Keywords: IPMNs; Intraductal Papillary Mucinous Neoplasms
MeSH Terms: interventions — Sensitivity and Specificity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Sensitivity and specificity of risk factors for degeneration of IPMNs — Measurement of high-grade dysplasia or invasive cancer on the histological analysis of the surgical specimen

SUMMARY:
Cystic lesions of the pancreas are frequent with a risk of degeneration into adenocarcinoma with pejorative prognosis.

IPMNs require characterization to clarify their potential for degeneration. Clinical and morphological risk factors for degeneration determine the monitoring rate and the indication for pancreatic surgery.

Pancreatic surgery remains invasive with high morbidity and mortality rates.

DETAILED DESCRIPTION:
This is a monoservice and monocentric retrospective study at the Nancy CHRU. We will study the risk factors for IPMNs degeneration in order to determine the most sensitive and specific.

To do this, we will use high-grade dysplasia or invasive cancer on the histological analysis of surgical specimens as the primary endpoint.

The study population will be patients with Branch Duct, Main Duct or mixed IPMNs operated at the Nancy CHRU between September 2009 and October 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Branch Duct, Main Duct or mixed IPMNs operated at the Nancy CHRU between September 2009 and October 2021, adults and without legal protection measures

Exclusion Criteria:

* IPMNs not operated
* Pancreatic cancer without IPMNs
* Patients whose state of health contraindicates pancreatic surgery
* Non-adult patient
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Branch Duct, Main Duct or mixed IPMNs operated at the Nancy CHRU between September 2009 and October 2021
Sampling Method: Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
High-grade dysplasia or invasive cancer | 12 years
  High-grade dysplasia or invasive cancer on histological analysis of the surgical specimen

CONTACTS AND LOCATIONS:
Overall Officials: Jean Baptiste JC CHEVAUX, Principal Investigator — Centre Hospitalier Regional Universitaire de Nancy
Locations (1):
- Jean-Baptiste CHEVAUX, Nancy, France

IPD SHARING:
Plan to Share IPD: No